CLINICAL TRIAL: NCT06504836
Title: Effects of Kinematic Biofeedback on Gait Quality in People With Stroke
Brief Title: Kinematic Biofeedback on Gait Quality in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112205AF1
Record Dates: First submitted 2024-06-30; First posted 2024-07-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Biofeedback; Gait symmetry; Gait variability
MeSH Terms: conditions — Stroke | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait training with biofeedback group (Experimental): The intervention is a single 60-minute session.
  Interventions: Other: Gait training with biofeedback
- Gait training without biofeedback group (Active Comparator): The intervention is a single 60-minute session.
  Interventions: Other: Gait training without biofeedback

INTERVENTIONS:
Other: Gait training with biofeedback — Gait training include treadmill and overground walking. The biofeedback device system will provide real-time feedback on hip extension angles.
  Arms: Gait training with biofeedback group
Other: Gait training without biofeedback — Gait training include treadmill and overground walking.
  Arms: Gait training without biofeedback group

SUMMARY:
Walking disorder is the most common and concerning issue for individuals with stroke. Previous studies have often used improvements in walking speed and distance as reference indicators for the advancement of gait performance in individuals with stroke. However, for individuals with chronic stroke, considering gait symmetry and variability to enhance gait quality as the primary intervention target may be more crucial. According to a literature review, it can be inferred that the application of biofeedback to detect gait quality may be an effective approach to improve gait symmetry and variability in individuals with stroke. However, there is still insufficient research evidence on this issue. Therefore, this study aims to investigate the effects of a kinematic biofeedback device system, which detects hip joint angles, on gait quality in individuals with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Stroke onset time ≥ 6 months
* Functional Ambulation Category ≥3
* Passive range of motion of affected hip extension is at least 10 degrees
* Mini-Mental State Measurement score ≥ 24 points

Exclusion Criteria:

* Modified Ashworth Scale of affected ankle plantar flexors ≥ 2
* Muscle strength of affected ankle plantar flexors via Manual Muscle Testing ≤ 1
* Uncorrected auditory impairment
* Severe cardiovascular disease or uncontrolled hypertension
* Other orthopedic diseases that may affect walking ability
* Other neurological disease except stroke

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait symmetry | 1 day
  Using GAITRite system to measure the symmetry of spatiotemporal parameters, including step length, step width, single support time, and double support time. Calculate the gait symmetry using following formula:
  Gait symmetry = affected side/ unaffected side.
Gait variability | 1 day
  Using GAITRite system to measure the coefficient of variation (CV). The mean and standard deviation will be used to calculate the coefficient of variation (CV).
  CV = standard deviation / mean * 100%

SECONDARY OUTCOMES:
Propulsive force | 1 day
  Using Force plate to measure the ground reaction force

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan